CLINICAL TRIAL: NCT00422851
Title: Gas Supply, Demand and Middle Ear Gas Balance: Specific Aim 3c
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, J. Douglas Swarts, Associate Professor, University of Pittsburgh
Other Study IDs: 0609093; NIH P50DC007667
Record Dates: First submitted 2007-01-12; First posted 2007-01-17 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Healthy
Keywords: otitis; gas diffusion; Eustachian tube; tympanic membrane
MeSH Terms: conditions — Otitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Normal tympanic membrane
- 2: tympanosclerosis
- 3: dimeric (atrophic)

SUMMARY:
This study will determine if gas can pass between the environment and the middle ear by way of the eardrum. This route of gas exchange was observed in animals but has not been studied in humans. If gas exchange across the eardrum is documented and the rate is sufficiently high, this can help explain certain past observations such as why middle ear pressure does not change very much in some children and adults when they have a cold or flu. The investigators also expect that the rate of gas exchange across the eardrum will depend on whether or not the eardrum has scarred or abnormally thin regions.

DETAILED DESCRIPTION:
Middle-ear (ME) pressure is a measure of the number of contained gas moles, and processes that addd or remove gas moles from the relatively fixed volume ME cavity change its pressure. Experimental results from animal studies document significant gas exchange across the tympanic membrane and if confirmed for humans may explain some of the paradoxical findings for children with poor Eustachian tube function such as the preservation of an aerated ME when the normal routes of gas supply are disrupted. This study measures the rates of reactive and inert gas exchange across the adult tympanic membrane with and without structural abnormalities and determines if these transfers are purely diffusive phenomena. The resulting data will be used to develop species-specific rate-constants that will be used as parameters in modeling ME pressure regulation.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old
* at least one intact and effusion-free middle ear

Exclusion Criteria:

* bilateral otitis media
* unable to remain relaxed and quiet for up to 2 hours

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults 18-50 years old with at least one intact and effusion-free middle ear
Sampling Method: Probability Sample
Enrollment: 45
Dates: Start 2007-06; Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Doyle, PhD, Principal Investigator — University of Pittsburgh; J. Douglas Swarts, PhD, Study Director — University of Pittsburgh
Locations (1):
- ENT Research Center Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States